CLINICAL TRIAL: NCT04883580
Title: A Prospective, Multicenter, Non Inferiority, Randomized Controlled Clinical Trial to Evaluate the Safety and Efficacy of Pedicle Screw Fixation Assisted by Orthopedic Surgical Navigation System
Brief Title: Navigation and Positioning System for Orthopedic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanjing Tuodao Medical Technology Co., Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-MD-100
Record Dates: First submitted 2021-05-07; First posted 2021-05-12 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Pedicle Screw Fixation of Spine
MeSH Terms: interventions — Orthopedic Procedures

STUDY DESIGN:
Intervention Model Description: NS100
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental)
  Interventions: Device: Navigation and Positioning System for Orthopedic Surgeries
- control group (Active Comparator)
  Interventions: Device: Navigation and Positioning System for Orthopedic Surgeries

INTERVENTIONS:
Device: Navigation and Positioning System for Orthopedic Surgeries — Experimental group: orthopedic surgery navigation system (Tuodao) assisted pedicle screw fixation
  Control group: orthopedic surgery navigation system (tianzhihang) assisted pedicle screw fixation

SUMMARY:
This clinical trial is a prospective, multicenter, non inferiority, randomized controlled trial. We plan to include 112 subjects in China and randomly assign them to the experimental group and the control group according to the ratio of 1:1. The experimental group used the orthopedic surgery navigation and positioning system produced by Nanjing Tuodao Medical Technology Co., Ltd., while the control group used the orthopedic surgery navigation and positioning system produced by Beijing tianzhihang Medical Technology Co., Ltd. Taking the position deviation of Kirschner wire as the main evaluation index, it was proved that the test instrument was not inferior to the control instrument. The test data shall be submitted to the State Drug Administration for approval of the marketing license of the test device

ELIGIBILITY:
Inclusion Criteria:

1. They were 18-75 years old;
2. From thoracic vertebrae to lumbar vertebrae, pedicle screw fixation is needed;
3. Signed informed consent, willing to receive treatment and follow-up according to the requirements of the trial protocol.

Exclusion Criteria:

1. Patients with pedicle deformity.
2. Patients with severe osteoporosis.
3. Patients with spinal tumor or tuberculosis.
4. Patients with abnormal liver function (alanine aminotransferase, aspartate aminotransferase values > 3 times of the upper limit of the normal range) and abnormal renal function (creatinine values > 3 times of the upper limit of the normal range).
5. Patients with abnormal coagulation function (prothrombin time, activated partial thromboplastin time > 1.5 times of the upper limit of normal range).
6. Pregnant or lactating women.
7. Patients with mental disorders.
8. The investigators evaluated patients who were not suitable for pedicle screw fixation.
9. Patients who are participating in clinical trials of any other device or drug.
10. Poor compliance, difficult to cooperate with patients who complete treatment and follow-up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2021-05-28 (Estimated); Primary Completion 2022-05-28 (Estimated); Study Completion 2022-05-28 (Estimated)

PRIMARY OUTCOMES:
Deviation of the position of Kirschner needle | Immediately after operation
  Comparing the actual placement position of Kirschner wire with the planned position of C-arm 3D scanning, the average deviation of the entry point and the insertion point was the position deviation of Kirschner wire

SECONDARY OUTCOMES:
Excellent and good rate of pedicle screw placement | Discharge or 7 days after surgery, whichever comes first
  Gertzbein Robbins classification criteria: whether there is cortical penetration in the lateral, medial, cephalic and caudal directions of pedicle screws (A: no cortical invasion; B: no cortical invasion); B: Cortical penetration was less than 2 mm; C: 2mm ≤ cortical penetration < 4mm; D: 4mm ≤ 6 mm; E: Cortical penetration ≥ 6 mm)
Entry point deviation | Immediately after operation
  The space distance between the entrance point of the planned position of the passage and the axis of the actual placement position of the Kirschner wire
Dead center deviation | Immediately after operation
  The space distance between the end point of the planned position of the passage and the axis of the actual placement position of the Kirschner wire
Angle deviation of axial plane | Immediately after operation
  The minimum angle between the planned position of the passage and the projection position of the Kirschner wire on the axial plane
Angular deviation of sagittal plane | Immediately after operation
  The minimum angle between the planned position of the passage and the projection position of the Kirschner wire on the sagittal plane
Spatial angle deviation | Immediately after operation
  The minimum angle between the planned position of the passage and the actual position of the Kirschner wire in space
Operation time | Immediately after operation
  The time from the beginning of registration to the end of the nail placement in the navigation and positioning system of orthopedic surgery
Incidence of re nailing | Immediately after operation
Incidence of conversion to manual nail placement | Immediately after operation
apparatus Success rate | Immediately after operation
  Instrument success refers to that during the operation, the operator completes the operation channel planning based on the three-dimensional scanning image data of the C-arm, and the orthopedic surgery navigation and positioning system makes the manipulator move to the position specified in the operation planning under the monitoring of the operator, without instrument defects
Technical success rate | Immediately after operation
  Technical success refers to the successful insertion of Kirschner wire along the guider and sleeve during the operation without re insertion or changing to manual insertion
Success rate of operation | Immediately after operation
  The success of operation refers to the success of instruments and techniques in the operation without serious complications
Incidence of device defects | Immediately after operation
  Device defect refers to the unreasonable risk of medical devices that may endanger human health and life safety in normal use, such as label error, quality problem, fault, etc
Incidence of severe surgical complications | Discharge or 7 days after surgery, whichever comes first
  Severe complications included nerve root injury, vascular injury, spinal cord injury, visceral injury and pedicle fracture
Incidence of adverse events and serious adverse events | Discharge or 7 days after surgery, whichever comes first

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tian W, Liu Y, Zheng S, Lv Y. Accuracy of lower cervical pedicle screw placement with assistance of distinct navigation systems: a human cadaveric study. Eur Spine J. 2013 Jan;22(1):148-55. doi: 10.1007/s00586-012-2494-6. Epub 2012 Sep 18. PMID 22987158
- [Result] Tian NF, Huang QS, Zhou P, Zhou Y, Wu RK, Lou Y, Xu HZ. Pedicle screw insertion accuracy with different assisted methods: a systematic review and meta-analysis of comparative studies. Eur Spine J. 2011 Jun;20(6):846-59. doi: 10.1007/s00586-010-1577-5. Epub 2010 Sep 23. PMID 20862593
- [Result] Devito DP, Kaplan L, Dietl R, Pfeiffer M, Horne D, Silberstein B, Hardenbrook M, Kiriyanthan G, Barzilay Y, Bruskin A, Sackerer D, Alexandrovsky V, Stuer C, Burger R, Maeurer J, Donald GD, Schoenmayr R, Friedlander A, Knoller N, Schmieder K, Pechlivanis I, Kim IS, Meyer B, Shoham M. Clinical acceptance and accuracy assessment of spinal implants guided with SpineAssist surgical robot: retrospective study. Spine (Phila Pa 1976). 2010 Nov 15;35(24):2109-15. doi: 10.1097/BRS.0b013e3181d323ab. PMID 21079498
- [Result] Burch S. Surgical complications of spinal deformity surgery. Neurosurg Clin N Am. 2007 Apr;18(2):385-92. doi: 10.1016/j.nec.2007.02.007. PMID 17556141
- [Result] Holly LT, Foley KT. Three-dimensional fluoroscopy-guided percutaneous thoracolumbar pedicle screw placement. Technical note. J Neurosurg. 2003 Oct;99(3 Suppl):324-9. doi: 10.3171/spi.2003.99.3.0324. PMID 14563154
- [Result] Kosmopoulos V, Schizas C. Pedicle screw placement accuracy: a meta-analysis. Spine (Phila Pa 1976). 2007 Feb 1;32(3):E111-20. doi: 10.1097/01.brs.0000254048.79024.8b. PMID 17268254
- [Result] Klein SA, Glassman SD, Dimar JR 2nd, Voor MJ. Evaluation of the fixation and strength of a "rescue" revision pedicle screw. J Spinal Disord Tech. 2002 Apr;15(2):100-4. doi: 10.1097/00024720-200204000-00002. PMID 11927817
- [Result] Tan SH, Teo EC, Chua HC. Quantitative three-dimensional anatomy of cervical, thoracic and lumbar vertebrae of Chinese Singaporeans. Eur Spine J. 2004 Mar;13(2):137-46. doi: 10.1007/s00586-003-0586-z. Epub 2003 Dec 12. PMID 14673715
- [Result] Laine T, Lund T, Ylikoski M, Lohikoski J, Schlenzka D. Accuracy of pedicle screw insertion with and without computer assistance: a randomised controlled clinical study in 100 consecutive patients. Eur Spine J. 2000 Jun;9(3):235-40. doi: 10.1007/s005860000146. PMID 10905443
- [Result] Holly LT, Foley KT. Intraoperative spinal navigation. Spine (Phila Pa 1976). 2003 Aug 1;28(15 Suppl):S54-61. doi: 10.1097/01.BRS.0000076899.78522.D9. PMID 12897475
- [Result] Mendelsohn D, Strelzow J, Dea N, Ford NL, Batke J, Pennington A, Yang K, Ailon T, Boyd M, Dvorak M, Kwon B, Paquette S, Fisher C, Street J. Patient and surgeon radiation exposure during spinal instrumentation using intraoperative computed tomography-based navigation. Spine J. 2016 Mar;16(3):343-54. doi: 10.1016/j.spinee.2015.11.020. Epub 2015 Dec 10. PMID 26686604
- [Result] Solomiichuk V, Fleischhammer J, Molliqaj G, Warda J, Alaid A, von Eckardstein K, Schaller K, Tessitore E, Rohde V, Schatlo B. Robotic versus fluoroscopy-guided pedicle screw insertion for metastatic spinal disease: a matched-cohort comparison. Neurosurg Focus. 2017 May;42(5):E13. doi: 10.3171/2017.3.FOCUS1710. PMID 28463620